CLINICAL TRIAL: NCT07284823
Title: Safety and Usability of the Cionic Neural Sleeve for Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cionic, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Webster, Clinical Operations Manager, Cionic, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIONIC-08-001
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cionic Neural Sleeve NS-200 (Experimental): Participants will wear the device during the study and receive stimulation assistance during walking.
  Interventions: Device: Cionic Neural Sleeve Multistim System

INTERVENTIONS:
Device: Cionic Neural Sleeve Multistim System — The sleeve assists participants during physical activity by delivering electrical stimulation that helps contract the necessary muscles at the correct time to improve movement.

SUMMARY:
This research will investigate the safety and usability of the Cionic Neural Sleeve Multistim System for Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported gait impairment
* Have access to a smartphone with iOS or Android operating system with Bluetooth capabilities and internet connection
* Ability to walk with or without an assistive device for up to 1 minute
* Leg measurements within sizing range of the Cionic Neural Sleeve

Exclusion Criteria:

* Daily occurrence of falls
* Implanted demand-type cardiac pacemaker or defibrillator
* Malignant tumor or existing thrombosis in the leg
* Fracture or dislocation in the leg that could be adversely affected by motion from stimulation

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Able to Independently Exit a Stimulation Program Using the Cionic Neural Sleeve | Day 0, Week 6, Week 12
  Participants' ability to independently exit (terminate) an active stimulation program on the Cionic Neural Sleeve will be assessed during study visits. Independence is defined as successful completion of the task without verbal cueing or physical assistance from study staff. Study staff will document whether the participant is able to exit the program independently (yes/no) at each visit.
Number of Participants Able to Independently Test Stimulation Using the Cionic Neural Sleeve | Day 0, Week 6, Week 12
  Participants' ability to independently initiate and test stimulation on the Cionic Neural Sleeve will be assessed during study visits. Successful task completion is defined as the participant correctly activating stimulation and confirming perception of stimulation without assistance. Study staff will document successful independent testing (yes/no).
Number of Participants Able to Independently Calibrate the Cionic Neural Sleeve System | Day 0, Week 6, Week 12
  Participants' ability to independently complete device calibration of the Cionic Neural Sleeve system will be assessed during study visits. Calibration is defined as completion of the device-guided calibration procedure without verbal or physical assistance. Study staff will document successful independent calibration (yes/no).
Safety of the Cionic Neural Sleeve | Day 0, Week 6, Week 12
  To understand the device's safety profile and potential side effects, researchers will record any adverse events during their home use.

OTHER OUTCOMES:
Qualitative Feedback on Stimulation Timing | Day 0, Week 6, Month 3
  Qualitative feedback regarding stimulation timing during gait will be collected every 6 weeks using structured interviews. Data will be used to assess user experience and perceived synchronization between stimulation delivery and functional movement.
Usability of the Cionic Neural Sleeve | Week 12
  Usability of the Cionic Neural Sleeve will be evaluated using the 10-item System Usability Scale with total scores ranging from 0 to 100. Scores greater than or equal to 68 indicate above-average usability.
Impact of the Cionic Neural Sleeve | Day 0, Week 6, Week 12
  The Timed Up and Go (TUG) test will be used to assess functional mobility. Participants are instructed to stand up from a chair, walk 3 meters, turn around, return to the chair, and sit down. The total time to complete the task is recorded in seconds, with shorter times indicating better mobility. A minimum clinically important difference (MCID) of 0.77 seconds will be used to interpret meaningful change in performance over time.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Adapt Movement, Carlsbad, California
  - CIONIC, San Francisco, California

IPD SHARING:
Plan to Share IPD: No